CLINICAL TRIAL: NCT01563692
Title: Analysis of the Immune Response to Respiratory Syncytial Virus (RSV) Infection in Health Care Personnel
Brief Title: Immune Response to Respiratory Syncytial Virus (RSV) in Health Care Workers
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: ReiThera Srl (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011/08
Record Dates: First submitted 2011-12-05; First posted 2012-03-27 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: RSV; Immune response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The humoral and cellular immune response to RSV exposure. To characterise these further some analysis of HLA typing my occur.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Paediatric health care workers: NHS members of staff who regularly care for children admitted with RSV infections, and who therefore have a higher rate of exposure.
- Non-paediatric health care workers: This is a comparator group made up of healthy adults who do not work in an occupation or have other risk factors for higher exposure to RSV.

SUMMARY:
Respiratory Syncytial Virus (RSV) is a human restricted pathogen and is the single most important cause of severe respiratory illness in infants and young children, a major cause of infantile bronchiolitis and is the most frequent cause of hospitalization of infants and young children in industrialized countries. Severe RSV infection early in life is associated with an increased risk of subsequent recurrent wheezing and asthma. There are few population-based estimates of the incidence of RSV disease from developing countries, but the existing data clearly indicates that the virus accounts for a high proportion of Acute Respiratory Infections (ARI) in children. Studies in Brazil, Colombia and Thailand suggest that RSV causes 20-30% of ARI cases in children from 1-4 years of age, a proportion similar to that in industrialized countries, and WHO has estimated the global RSV disease burden at 64 million cases and 160 000 deaths every year. RSV also causes severe disease in elderly and immune-compromised adults, and the burden of RSV disease in the elderly is comparable to that of seasonal influenza. The economic impact of RSV-related disease in adults estimated to be greater than that of influenza in relation to numbers of days lost from work.

The development of a safe and effective vaccine against RSV would benefit greatly from data on the immune responses in healthy adults naturally exposed to the virus. RSV infection has been shown to increase and induce short-lived circulating antibody secreting cells and produce an increase in the RSV specific antibody titres but very limited data is available on the cellular immune responses induced by RSV during natural infection in healthy adults. The existence of cell mediated immune response against RSV in humans has been described but characterization of this response remains poor and simultaneous analysis of several immunological parameters have not been attempted in an RSV exposed population before.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study and comply with study requirements
* Male or Female, aged from 18 to 60 in healthy status.
* Working on a paediatric ward which admits acute medical paediatric admissions during the RSV season (Group 1 only).

Exclusion Criteria:

* History of any immunodeficiency or immunological disorder which could affect the acquisition of RSV responses.
* Use of immunosuppressive medications such as steroids.
* Working on an NHS ward or in close contact with populations at higher risk of RSV transmission (e.g. nursery workers, care home workers, parents of young children) during the RSV season (Group 2 only).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy health care personnel working in a pediatric ward and healthy volunteers from non-NHS staff
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Immune response to natural RSV exposure | July 2012 (up to 4 months)
  To assess the induction of cellular responses and antibodies following natural exposure to RSV

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, PhD, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, United Kingdom

REFERENCES:
- [Derived] Green CA, Sande CJ, de Lara C, Thompson AJ, Silva-Reyes L, Napolitano F, Pierantoni A, Capone S, Vitelli A, Klenerman P, Pollard AJ. Humoral and cellular immunity to RSV in infants, children and adults. Vaccine. 2018 Oct 1;36(41):6183-6190. doi: 10.1016/j.vaccine.2018.08.056. Epub 2018 Aug 31. PMID 30177258